CLINICAL TRIAL: NCT06463938
Title: A Clinical Study to Evaluate the Effectiveness of Casein Phosphopeptide, Amorphous Calcium Phosphate Paste (CPP-ACP) Used Alone or in Combination With Lasotronix (Diode Laser) to Treat Dentin Hypersensitivity
Brief Title: A Clinical Trial to Compare Lasotronix Alone or in Combination With CPP-ACP to Treat DH
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Dow University of Health Sciences (Other)
Responsible Party: Principal Investigator, Sanam Faheem, Senior Lecturer, Dow University of Health Sciences
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: Dow
Record Dates: First submitted 2024-06-11; First posted 2024-06-18 (Actual); Last update posted 2024-07-26 (Actual); Status verified 2024-07

CONDITIONS: Dentin Sensitivity; Hypersensitivity; Cervical Lesion
Keywords: Dentin Sensitivity; Lasotronix; Diode laser
MeSH Terms: conditions — Dentin Sensitivity; Hypersensitivity | interventions — Ointments; Control Groups

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Active Comparator (Active Comparator): would include patients (n=30) who will be given CPP-ACP paste application only
  Interventions: Other: Active comparator
- Experimental (Experimental): would consist of patients (n=30) who will be given diode laser therapy only
  Interventions: Device: Experimental group
- Combination (Other): would include patients (n=30) who will be given a combination of CPP-ACP paste & Laser therapy.
  Interventions: Combination Product: Combination of laser and paste
- Control (Other): would be a control group
  Interventions: Behavioral: Control group

INTERVENTIONS:
Other: Active comparator — CPP-ACP paste will be applied on exposed area
  Arms: Active Comparator
Device: Experimental group — Lasotronix will be applied following its protocol
  Arms: Experimental
Combination Product: Combination of laser and paste — This group will receive the combination of above two treatments
  Arms: Combination
Behavioral: Control group — this will be a control group
  Arms: Control

SUMMARY:
Dentin hypersensitivity (DH) is defined as sharp pain of a shorter duration arise from exposed dentin in response to several chemicals and thermal or tactile stimuli that cannot be ascribed to other dental defects". DH has a prevalence rate ranging from 1.3% to 92.1%, commonly affecting old ages. The use of laser has opened new dimensions in the treatment of DH. To the author's knowledge, not much research work has been conducted using LASOTRONIX as a treatment modality with CPP-ACP. Therefore, this research aims to determine the effectiveness of Casein phospho peptide paste (CPP-ACP) used alone or combined with a diode laser (LASOTRONIX).

DETAILED DESCRIPTION:
DH has a prevalence rate ranging from 1.3% to 92.1%, commonly affecting old ages, and the frequency of DH in patients suffering from periodontal disease is 3-57%. Pakistan has reported prevalence from different cities, with 36.4% from Karachi and 22% from Lahore.

The use of laser has opened new dimensions in the treatment of DH. Theories that support laser therapy explain that irradiation blocks the pain in dentinal tubules by melting and recrystallization of dentin or by tertiary dentine production or evaporation of dentinal fluid. Considering the oral soft tissues which contain high amounts of water, Lasotronix SMARTm laser diodes have been carefully designed to show their high transmission. The 635nm wavelength is optimal for activating tolonium chloride dye for photo-activated chemo therapy, eliminating all bacteria and biofilms without any side effects. 200 mW power provides safe cold bio stimulation and photo disinfection within a reasonably short therapy time. Application of Sodium fluoride (NaF) has also been indicated for hypersensitivity pains. Its application in the form of gel occludes the tubule by calcium fluoride precipitation. Agents like potassium nitrate also have promising effects, which increase the concentration of potassium ions in nerve endings and alter the nerve action potential in conducting the sensory stimuli.

Recently DH treatment has been conducted with different types of laser with different wavelengths, either alone or in combination with desensitizing agents and varnishes and has revealed effective results. To the author's knowledge, not much research work has been conducted using LASOTRONIX as a treatment modality with CPP-ACP. Therefore, this research aims to determine the effectiveness of Casein phospho peptide paste (CPP-ACP) used alone or combined with a diode laser (LASOTRONIX).

ELIGIBILITY:
Inclusion criteria:

* Patients of either gender, with ages between 25-65 years
* should have at least more than one hypersensitive and vital tooth without any carious lesion or defective restoration

Exclusion criteria:

* History of desensitizing therapy on the affected tooth/teeth in last six months (use of desensitizing toothpaste)
* use of antibiotics /analgesic/anti-inflammatory drugs
* history of smoking
* pregnancy
* those who are not willing to participate or give follow-ups

Ages: 25 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 120 (Estimated)
Dates: Start 2024-05-12 (Actual); Primary Completion 2024-08-10 (Estimated); Study Completion 2024-10-10 (Estimated)

PRIMARY OUTCOMES:
treatment of dentin hypersensitivity | 0-3 moths
  VAS Visual analogue scale will be used to determine the efficacy of different treatment methods.

CONTACTS AND LOCATIONS:
Locations (1):
- Dr Sanam Faheem, Karachi, Sindh, Pakistan

IPD SHARING:
Plan to Share IPD: Yes